CLINICAL TRIAL: NCT00475423
Title: An Open Label Study of a Fixed Dose Regimen of MabThera on Overall Response Rate in Patients With Refractory, Relapsing or Chronic Idiopathic Thrombocytopenic Purpura.
Brief Title: A Study of MabThera (Rituximab) in Patients With Idiopathic Thrombocytopenic Purpura.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20948
Record Dates: First submitted 2007-05-17; First posted 2007-05-21 (Estimated); Results first posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Idiopathic Thrombocytopenic Purpura
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: rituximab [MabThera/Rituxan] — 1000mg iv on days 1 and 15

SUMMARY:
This single arm study will evaluate the efficacy and safety of MabThera monotherapy in patients with refractory, relapsing or chronic idiopathic thrombocytopenic purpura (ITP). Patients will receive infusions of MabThera 1000mg i.v. on days 1 and 15. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* refractory, relapsing or chronic idiopathic thrombocytopenic purpura;
* stable therapy during 3 weeks prior to study entry.

Exclusion Criteria:

* newly diagnosed ITP (<6 weeks);
* prior treatment with MabThera;
* active bleeding requiring platelet transfusion within 7 days prior to entry into study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-05; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (11):
- Australia (11):
  - Adelaide, New South Wales
  - Gosford, New South Wales
  - Randwick, New South Wales
  - Sydney, New South Wales
  - Westmead, New South Wales
  - Woolloongabba, Queensland
  - Adelaide, South Australia
  - Frankston, Victoria
  - Malvern, Victoria
  - Melbourne, Victoria
  - Parkville, Victoria

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Participants received rituximab 1000 milligrams (mg) intravenously (IV) on Days 1 and 15.
Period: Overall Study
Arm/Group | Rituximab
Started | 122
Completed | 90
Not Completed | 32
Not completed — Protocol Violation | 5
Not completed — Adverse Event | 4
Not completed — Withdrawal by Subject | 6
Not completed — Lack of Efficacy | 8
Not completed — Death | 1
Not completed — Reason not specified | 1
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Population: Safety population: all participants who received at least one dose of study medication and for whom follow-up safety information was available.
Groups:
- Rituximab: Participants received rituximab 1000 mg IV on Days 1 and 15.
Arm/Group | Rituximab
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.5 (18.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Complete Hematological Response (CR) or Confirmed Partial Hematological Response (PR)
Description: Percentage of participants with an overall response at Week 8 achieving a CR or PR as evaluated by platelets, new or increased Idiopathic Thrombocytopenic Purpura (ITP)-related treatments and corticosteroids given for Adverse Events (AEs). CR was defined as a platelet count of greater than (>) 150x10^9/ liters (L) over at least 2 consecutive measurements at least 2 weeks apart, but no more than 60 days apart, with no increase in concomitant ITP therapy or initiation of new ITP therapy. PR was defined as platelet count of >50x10^9/L over at least 2 consecutive measurements at least <2 weeks apart, but no more than 60 days apart, with no increase in concomitant ITP therapy or initiation of new ITP therapy. Overall response rate (participants who achieved CR or confirmed PR) was evaluated using platelets, new or increased ITP related treatments, and corticosteroids given for AEs.
Time Frame: Week 8
Population: Intent-to-Treat Replaced (ITTR) Population: participants who received at least 1 dose of study medication, excluded those lost to follow-up before completing treatment (reasons other than disease progression/toxicity) and/or those without documented platelet count of less than or equal to (≤)50x10^9/L within 7 days prior to 1st rituximab infusion.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rituximab 1000 mg: Participants received rituximab 1000 mg IV on Days 1 and 15.
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
percentage of participants | 43.5 [34.0 to 53.4]

2. Secondary Outcome: Percentage of Participants With Hematological CR, PR, or Minor Response (MR)
Description: Percentage of participants with CR, PR, and MR at Week 8 as evaluated by platelet count where CR is greater than or equal to (≥)150x10^9/L, PR ≥ 50x10^9/L, MR equals (=) 30x10^9/L over 2 consecutive measurements at least 2 weeks apart but no more than 60 days apart with no increase in concomitant therapy or initiation of new ITP therapy.
Time Frame: Week 8
Population: ITTR Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
percentage of participants
  CR | 9.3 [4.5 to 16.4]
  PR | 34.3 [25.4 to 44.0]
  MR | 17.6 [10.9 to 26.1]

3. Secondary Outcome: Percentage of Participants Who Achieved CR
Description: CR was defined as platelet counts >150x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, and with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Week 52
Population: ITTR Population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
percentage of participants | 27.8

4. Secondary Outcome: Time to CR
Description: Time to CR was defined as the time from the first infusion to the first date on which CR was achieved. CR was defined as platelet counts >150x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, and with no increase in concomitant ITP therapy or initiation of new ITP therapy. Participants without an event were censored at the date of last assessment.
Time Frame: Baseline to Week 52
Population: ITTR Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
days | NA [305.0 to NA] — Median time to CR and upper limit of the 95% confidence interval could not determined due to an insufficient number of events.

5. Secondary Outcome: Percentage of Participants Who Achieved PR
Description: PR was defined as platelet counts >50x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Week 52
Population: ITTR Population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
percentage of participants | 56.5

6. Secondary Outcome: Time to PR
Description: Time to response was defined as the time from the first infusion to the first date on which PR was achieved. PR was defined as platelet counts > 50x10^9/L over ≥ 2 consecutive measurements ≥ 2 weeks apart, but no more than 60 days apart, with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Baseline to Week 52
Population: ITTR Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
days | 53.0 [36.0 to 152.0]

7. Secondary Outcome: Percentage of Participants Who Achieved MR
Description: MR was defined as participants registered with chronic ITP with a platelet count of >30x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, with a 50 to 100% reduction in the dose intensity of concomitant ITP therapy compared with that at screening, and with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Week 52
Population: ITTR Population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
percentage of participants | 71.3

8. Secondary Outcome: Time to MR
Description: Time to response was defined as the time from the first infusion to the first date on which MR was achieved. MR was defined as participants registered with chronic ITP with a platelet count of >30x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, with a 50 percent (%) to 100% reduction in the dose intensity of concomitant ITP therapy compared with that at screening, and with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Baseline to Week 52
Population: ITTR Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
days | 22.0 [8.0 to 30.0]

9. Secondary Outcome: Percentage of Participants With Continued CR From Week 8 to Week 52
Description: The number of participants with a durable CR assessed in CR responders whose responses were sustained from Week 8 through to the end of the study or withdrawal, irrespective of change of treatment. CR was defined as platelet counts >150x10^9/L over ≥2 consecutive measurements ≥ 2 weeks apart, but no more than 60 days apart, and with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Week 8 to Week 52
Population: ITTR Population; only participants with a CR at Week 8 were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 10
percentage of participants | 10

10. Secondary Outcome: Duration of CR in Participants With Continued CR From Week 8 Until Week 52
Description: Duration of response was assessed in all responders who reached Week 8 and was defined as the time from Week 8 to the end of CR, irrespective of change of treatment. CR was defined as platelet counts >150x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, and with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Week 8 to Week 52
Population: ITTR Population; only participants with a CR at Week 8 were included in the analysis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 10
days | NA [NA to NA] — Median and 95% confidence interval (CI) could not be calculated due an insufficient number of events.

11. Secondary Outcome: Duration of PR in Participants With Continued PR From Week 8 Until Week 52
Description: Duration of PR was assessed in all responders who reached Week 8 and was defined as the time from Week 8 to the end of PR, irrespective of change of treatment. PR was defined as platelet counts >50x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Week 8 to Week 52
Population: ITTR Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 47
days | 247.0 [219.0 to NA] — Upper limit of the 95% CI could not be calculated due to inadequate data.

12. Secondary Outcome: Duration of MR in Participants With Continued MR From Week 8 Until Week 52
Description: Duration of response was assessed in all responders who reached Week 8 and was defined as the time from Week 8 to the end of MR, irrespective of change of treatment. MR was defined as participants registered with ITP in relapse with a platelet count of > 30x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, with no increase in concomitant ITP therapy or initiation of new ITP therapy. Participants registered with chronic ITP with a platelet count of >30x10^9/L over ≥2 consecutive measurements ≥2 weeks apart, but no more than 60 days apart, with a 50% to 100% reduction in the dose intensity of concomitant ITP therapy compared with that at screening, and with no increase in concomitant ITP therapy or initiation of new ITP therapy.
Time Frame: Week 8 to Week 52
Population: ITTR Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 66
days | 256.0 [168.0 to NA] — Upper limit of 95% CI could not be calculated due to inadequate data.

13. Secondary Outcome: Time to Inititiation of New ITP Therapy - Percentage of Participants With an Event
Description: Percentage of participants with an event of initiation of new ITP therapy and/or increase in dose of existing ITP therapy, including date on which decision made in relation to splenectomy, from time of first treatment to Week 52.
Time Frame: Week 52
Population: ITTR Population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
percentage of participants | 50.0

14. Secondary Outcome: Time to Initiation of New ITP Therapy
Description: Median time in days to initiation of new ITP therapy and/or increase in dose of existing ITP therapy, including date on which decision made in relation to splenectomy, from time of first treatment to Week 52.
Time Frame: Baseline to Week 52
Population: ITTR Population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
days | 314.0 [215.0 to NA] — Upper limit of the 95% CI could not be calculated due to censored or missing data.

15. Secondary Outcome: Percentage of Therapeutic Responders
Description: Percentage of participants with a therapeutic response, defined as achieving CR, PR, or MR assessed at Week 26 and Week 52 or hematological response, defined as achieving CR, PR, or MR at Week 8. CR was defined as no platelet response or no reduction in the dose intensity of concomitant ITP therapy compared with that at screening. PR response was defined as at least a minor platelet response that enabled a 50% to 99% reduction in the dose intensity of concomitant ITP therapy compared with that at screening. MR was defined as at least a minor platelet response that enabled a 1% to 49% reduction in the dose intensity of concomitant ITP therapy compared with that at screening.
Time Frame: Week 26 and Week 52
Population: ITTR Population
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
percentage of participants
  Week 26 | 43.5
  Week 52 | 35.2

16. Secondary Outcome: Percentage of Participants With a Therapeutic Response
Description: Number of therapeutic responder participants by CR, PR, MR, or no response (NR) measured at Week 26 and Week 52. CR was defined as no platelet response or no reduction in the dose intensity of concomitant ITP therapy compared with that at screening. PR was defined as at least minor platelet response that enabled a 50% to 99% reduction in the dose intensity of concomitant ITP therapy compared with that at screening. MR was defined as at least minor platelet response that enabled a 1% to 49% reduction in the dose intensity of concomitant ITP therapy compared with that at screening.
Time Frame: Week 26 and Week 52
Population: ITTR Population
Measure: Number (95% Confidence Interval); unit: percentage participants
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 108
percentage participants
  Week 26: CR | 38.0 [28.8 to 47.8]
  Week 26: PR | 5.6 [2.1 to 11.7]
  Week 26: MR | 0.0 [0.0 to 3.4]
  Week 26: NR | 56.5 [46.6 to 66.0]
  Week 52: CR | 35.2 [26.2 to 45.0]
  Week 52: PR | 0.0 [0.0 to 3.4]
  Week 52: MR | 0.0 [0.0 to 3.4]
  Week 52: NR | 64.8 [55.0 to 73.8]

17. Secondary Outcome: Cluster of Differentiation 19 (CD19) B Cell Count
Description: Value of mean CD19+ B cell count at baseline. The standard reference range for CD19 is 0.05 to 0.35 x10^9/L.
Time Frame: Baseline, Weeks 1, 3, and 8, Follow-up Months 4, 6, 8, 10, and 12, and Last Day
Population: Safety Analysis Population; n (number) = number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 122
10^9 cells/L
  Baseline (n=84) | 0.27 (0.374)
  Week 1 (n=3) | 0.30 (0.251)
  Week 3 (n=96) | 0.01 (0.052)
  Week 8 (n=89) | 0.01 (0.033)
  Follow-up Month 4 (n=57) | 0.01 (0.029)
  Follow-up Month 6 (n=79) | 0.03 (0.041)
  Follow-up Month 8 (n=57) | 0.07 (0.085)
  Follow-up Month 10 (n=48) | 0.15 (0.315)
  Follow-up Month 12 (n=70) | 0.18 (0.289)
  Last Day (n=101) | 0.13 (0.252)

18. Secondary Outcome: Change From Baseline in CD19 B Cell Count
Description: Actual values of CD19+ mean B cell count assessed at Weeks 3 and 8, and Months 4, 6, 8, 10 and 12, and last day. The standard reference range for CD19 is 0.05 to 0.35 x10^9/L.
Time Frame: Weeks 3, 8 and Months 4, 6, 8, 10 and 12, and last day
Population: Safety Analysis Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Rituximab 1000 mg
Number analyzed (Participants) | 122
10^9 cells/L
  Week 3 (n=81) | -0.23 (0.290)
  Week 8 (n=75) | -0.27 (0.393)
  Follow-up Month 4 (n=47) | -0.21 (0.217)
  Follow-up Month 6 (n=63) | -0.23 (0.367)
  Follow-up Month 8 (n=44) | -0.22 (0.412)
  Follow-up Month 10 (n=39) | -0.08 (0.207)
  Follow-up Month 12 (n=55) | -0.06 (0.409)
  Last Day (n=84) | -0.13 (0.389)

ADVERSE EVENTS:
Time Frame: Up to Week 52
Arm/Group | Rituximab 1000 mg
Serious Adverse Events (participants affected / at risk) | 12/122
Other Adverse Events (participants affected / at risk) | 62/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg (N=122)
Asbestosis (Injury, poisoning and procedural complications) | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 1
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1
Streptococcal Bacteraemia (Infections and infestations) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Platelet Count Decreased (Investigations) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Stress (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab 1000 mg (N=122)
Nasopharyngitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 4
Respiratory tract infection (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Diarrhoea (Gastrointestinal disorders) | 5
Gingival bleeding (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Gastrointestinal pain (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Gingival pain (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Influenza like illness (General disorders) | 3
Pyrexia (General disorders) | 2
Chest pain (General disorders) | 1
Chills (General disorders) | 1
Ill-defined disorder (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 9
Fall (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 7
Dizziness (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 2
Cognitive disorder (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 5
Urticaria (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin pruritic (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2
Hot flush (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Ear haemorrhage (Ear and labyrinth disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Platelet count decreased (Investigations) | 2
Intraocular pressure increased (Investigations) | 1
Hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Serum sickness (Immune system disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Breast haematoma (Reproductive system and breast disorders) | 1
Eye pain (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Palpitation (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.